CLINICAL TRIAL: NCT06270433
Title: Efficacy and Safety of Toludesvenlafaxine Hydrochloride Sustained-release Tablets Versus Desvenlafaxine Succinate Sustained-release Tablets Targeting Anhedonia in Patients With Major Depression Disorder: a Multicentre, Open-label, Parallel-group, Randomised Controlled Trial
Brief Title: Efficacy and Safety of Toludesvenlafaxine Hydrochloride Sustained-release Tablets Versus Desvenlafaxine Succinate Sustained-release Tablets Targeting Anhedonia in Patients With Major Depression Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-KY142-01
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Anhedonia
MeSH Terms: conditions — Anhedonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toludesvenlafaxine hydrochloride sustained-release tablets treatment group (Experimental)
  Interventions: Drug: Toludesvenlafaxine hydrochloride sustained-release tablets
- Desvenlafaxine succinate sustained-release tablets treatment group (Active Comparator)
  Interventions: Drug: Desvenlafaxine succinate sustained-release tablets

INTERVENTIONS:
Drug: Toludesvenlafaxine hydrochloride sustained-release tablets — 80 mg or 120 mg or 160 mg orally once daily dosing for 8 weeks
  Arms: Toludesvenlafaxine hydrochloride sustained-release tablets treatment group
Drug: Desvenlafaxine succinate sustained-release tablets — 50 mg orally once daily dosing for 8 weeks
  Arms: Desvenlafaxine succinate sustained-release tablets treatment group

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of toludesvenlafaxine hydrochloride sustained-release tablets in the treatment of anhedonia in patients with major depression disorder compared to desvenlafaxine succinate sustained-release tablets, to provide evidence-based basis for clinical rational drug use.

DETAILED DESCRIPTION:
The study included 80 patients with major depression disorder (aged 18 to 65 years) who meet the diagnostic criteria for depression in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). Eligible patients were randomly assigned (1:1) to 8-week treatment with toludesvenlafaxine hydrochloride sustained-release tablets (n=40) or desvenlafaxine succinate sustained-release tablets(n=40), followed up at period of enrollment as baseline and at the end of 2th, 4th and 8th weeks. Adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meet the diagnostic criteria for major depression disorder in the Diagnostic and Statistical Manual of Manual Disorders, fifth Edition (DSM-5);
* Male or female aged ≥18 and ≤65 years;
* Subjects who have a Montgomery-Asberg Depression Rating Scale (MADRS) total score ≥24 points;
* Subjects who have a total score of Snaith-Hamilton Pleasure Scale (SHARPS) ≥3 points;
* Subjects voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

* Allergic or known to be allergic to toludesvenlafaxine hydrochloride sustained-release tablets and desvenlafaxine succinate sustained-release tablets;
* Subjects have a severe self-injury/clear suicide attempt or behavior; Scores on MADRS items factor 10 ≥4 points;
* Subjects who meet the diagnostic criteria for any other psychotic disorders (except for major depression disorder) in DSM-5, or those who have substance disorders or drug abuse within the past six months;
* Individuals with severe and unstable physical diseases such as cardiovascular disease, liver disease, kidney disease, blood disorders, and endocrine disorders;
* Hypertensive patients with poor blood pressure control (systolic blood pressure (SBP) ≥140 mmHg or diastolic blood pressure (DBP) ≥90 mmHg at screening);
* Total bilirubin (TBIL) values 1.5 times / alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 2 times / creatinine (Cr) 1.2 times higher than the upper limit of normal, or Thyroid-stimulating hormone (TSH) outside the normal range at screening;
* Electrocardiogram (ECG) abnormalities that are clinically significant at period of screening and that the investigator considers as inappropriate conditions for inclusion, such as QTc interval >450 ms in men and QTc interval >460 ms in female;
* Pregnant or lactating women, recent planned pregnancy and unable to ensure effective contraception during the period;
* Other conditions that the investigator considers the participant is not suitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Snaith-Hamilton Pleasure Scale (SHAPS) Total Score | Baseline and the end of week 8
  The SHAPS is a well-validated 14-item self-report questionnaire commonly used to assess anhedonia. Each item on the SHAPS is worded so that higher scores indicate greater pleasure capacity. A total score can be derived by summing the responses to each item. Each item is rated as either 0 or 1, for a total score between 0 and 14

SECONDARY OUTCOMES:
Snaith-Hamilton Pleasure Scale (SHAPS) Total Score | Baseline, the end of Week 2 and 4
  The SHAPS is a well-validated 14-item self-report questionnaire commonly used to assess anhedonia. Each item on the SHAPS is worded so that higher scores indicate greater pleasure capacity. A total score can be derived by summing the responses to each item. Each item is rated as either 0 or 1, for a total score between 0 and 14.
Snaith-Hamilton Pleasure Scale (SHAPS) Reductive Rate | The end of Week 2, 4 and 8
  SHAPS Reductive Rate(%) = (pre-treatment score - post-treatment score)/pre-treatment score ×100%.
Dimensional Anhedonia Rating Scale (DARS) Score | Baseline, the end of Week 2, 4 and 8
  DARS is a 17-item self-report questionnaire that is designed to assess anhedonia in major depressive disorder (MDD), and particularly to increase scale generalizability while maintaining specificity. Respondents provide their own examples of rewarding experiences across the domains of hobbies, social activities, food/drink, and sensory experience. Participants answer a set of standardized questions about desire, motivation, effort, and consummatory pleasure with a recall period of "right now" for the examples provided. The instrument is scored as a total sum of all items (range 0-68) with higher scores reflecting increased motivation, effort and pleasure (that is, less anhedonia).
Montgomery-Asberg Depression Rating Scale (MADRS) Score | Baseline, the end of Week 2, 4 and 8
  The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
17-item Hamilton Depression Rating Scale (HAM-D17) Score | Baseline, the end of Week 2, 4 and 8
  HAM-D17 has been the gold standard for the assessment of depression. The score needs to be based on clinical interviews, and the time frame of the assessment is usually the situation in the previous week. Most items use a 5-point scale of 0 to 4. The standard of each level is: 0 indicates none, 1 indicates mild, 2 indicates moderate, 3 indicates severe, and 4 indicates extremely severe. A few items adopt the 3-level scoring method with 0~2 points, and the grading standard is: 0 indicates none, 1 indicates mild to moderate and 2 indicates severe.
Sheehan Disability Scale (SDS) Score | Baseline, the end of Week 2, 4 and 8
  SDS is composed of three self-rating dimensions, which assess functional status in work, social life/leisure activities, and family life/family responsibilities. Each dimension is scored on a scale of 0 to 10, with 1 to 3 indicating mild impairment, 4 to 6 indicating moderate impairment, 7 to 9 indicating significant impairment, and 10 indicating extreme severity. The three dimensions can also be added together to reflect the overall functional deficiency. The score ranges from 0 to 30, with 0 indicating no damage and 30 indicating significant damage.
Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) Score | Baseline, the end of Week 2, 4 and 8
  Q-LES-Q-SF consists of 16 self-rated items. Each item is divided into five grades: 1 indicates very dissatisfied, 2 indicates dissatisfied, 3 indicates average, 4 indicates satisfied, and 5 indicates very satisfied. The higher the score, the better the happiness and quality of life satisfaction of the subjects. The first 14 items are used to generate an overall score, while the remaining 2 items are individual items that measure satisfaction and overall quality of life related to the study drug.

OTHER OUTCOMES:
Rating Scale for Side Effects (SERS) Score | The end of Week 2, 4 and 8
  All items in SERS adopt 4-level scoring method ranging from 0 to 3 points, and the standard of each item is as follows :0 indicates none, 1 indicates mild, 2 indicates moderate and 3 indicates severe. Two evaluation scales are required for each symptom. The first is the spontaneous reporting of patients when answering questions. The second is what the evaluator observed. The evaluator needs to systematically ask about each symptom.
Arizona Sexual Experience Scale (ASEX) Score | Baseline, the end of Week 2, 4 and 8
  ASEX is designed to assess aspects of psychotropic drug-induced sexual dysfunction: drive, arousal, penile erection/vaginal lubrication, ability to reach orgasm, and satisfaction from orgasm. The ASEX can be self- or clinician-administered. The 5 questions are rated using 6-point Likert-type scales with varying endpoints. Possible total scores range from 5 to 30, with the higher scores indicating more sexual dysfunction.
Count of red blood cell in blood | Baseline, the end of Week 8
  To analysis whether count of red blood cell in blood show any significant trend with time changes.
Count of white blood cell in blood | Baseline, the end of Week 8
  To analysis whether count of white blood cell in blood show any significant trend with time changes.
Count of platelet in blood | Baseline, the end of Week 8
  To analysis whether count of platelet in blood show any significant trend with time changes.
Concentration of hemoglobin in blood | Baseline, the end of Week 8
  To analysis whether concentration of hemoglobin in blood show any significant trend with time changes.
Concentration of alanine aminotransferase in blood | Baseline, the end of Week 8
  To analysis whether concentration of alanine aminotransferase in blood show any significant trend with time changes.
Concentration of aspartate aminotransferase in blood | Baseline, the end of Week 8
  To analysis whether concentration of aspartate aminotransferase in blood show any significant trend with time changes.
Concentration of gamma-glutamyltransferase in blood | Baseline, the end of Week 8
  To analysis whether concentration of gamma-glutamyltransferase in blood show any significant trend with time changes.
Concentration of blood glucose in blood | Baseline, the end of Week 8
  To analysis whether concentration of blood glucose in blood show any significant trend with time changes.
Concentration of serum creatinine in blood | Baseline, the end of Week 8
  To analysis whether concentration of serum creatinine in blood show any significant trend with time changes.
Concentration of urea in blood | Baseline, the end of Week 8
  To analysis whether concentration of urea in blood show any significant trend with time changes.
Concentration of total cholesterol in blood | Baseline, the end of Week 8
  To analysis whether concentration of total cholesterol in blood show any significant trend with time changes.
Concentration of high density lipoprotein in blood | Baseline, the end of Week 8
  To analysis whether concentration of high density lipoprotein in blood show any significant trend with time changes.
Concentration of low density lipoprotein in blood | Baseline, the end of Week 8
  To analysis whether concentration of low density lipoprotein in blood show any significant trend with time changes.
Concentration of triglyceride in blood | Baseline, the end of Week 8
  To analysis whether concentration of triglyceride in blood show any significant trend with time changes.
Concentration of thyroid-stimulating hormone in blood | Baseline, the end of Week 8
  To analysis whether concentration of thyroid-stimulating hormone in blood show any significant trend with time changes.
Concentration of protein in urine | Baseline, the end of Week 8
  To analysis whether concentration of protein in urine show any significant trend with time changes.
Concentration of sugar in urine | Baseline, the end of Week 8
  To analysis whether concentration of sugar in urine show any significant trend with time changes
Count of white blood cell in urine | Baseline, the end of Week 8
  To analysis whether count of white blood cell in urine show any significant trend with time changes.
Count of red blood cell in urine | Baseline, the end of Week 8
  To analysis whether count of red blood cell in urine show any significant trend with time changes.
ECG QT Interval | Baseline, the end of Week 8
  To analysis whether ECG QT Interval of participants show any significant trend with time changes.
Changes in weight | Baseline, the end of Week 2, 4 and 8
  To analysis whether weight of participants show any significant trend with time changes.
Changes in pulse | Baseline, the end of Week 2, 4 and 8
  To analysis whether pulse of participants show any significant trend with time changes.
Changes in both systolic and diastolic blood pressure | Baseline, the end of Week 2, 4 and 8
  To analysis whether blood pressure including systolic blood pressure and diastolic blood pressure of participants show any significant trend with time changes.
Changes in respiration rate | Baseline, the end of Week 2, 4 and 8
  To analysis whether respiration rate of participants show any significant trend with time changes.
Changes in armpit temperature | Baseline, the end of Week 2, 4 and 8
  To analysis whether armpit temperature of participants show any significant trend with time changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Brian Hospital, Nanjing, Jiangsu, China